CLINICAL TRIAL: NCT03904498
Title: COMT Inhibition as a Potential Therapeutic Target Among Individuals With Comorbid Alcohol Use Disorder and Attention-Deficit/Hyperactivity Disorder
Brief Title: COMT Inhibition Among Individuals With Comorbid AUD/ADHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-2335; R01AA026859 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Alcoholism; Attention Deficit Disorder with Hyperactivity | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tolcapone then Placebo (Experimental): Participants in this arm will receive tolcapone during the first medication period (1 capsule containing 200 mg tolcapone on study days 1 and 2; 3 capsules containing a total of 600 mg tolcapone on study days 3-8), and placebo during the second medication period (1 capsule on study days 1 and 2; 3 capsules on study days 3-8).
  Interventions: Drug: Tolcapone; Drug: Placebo
- Placebo then Tolcapone (Experimental): Participants in this arm will receive placebo during the first medication period (1 capsule on study days 1 and 2; 3 capsules on study days 3-8), and tolcapone during the second medication period (1 capsule containing 200 mg tolcapone on study days 1 and 2; 3 capsules containing a total of 600 mg tolcapone on study days 3-8).
  Interventions: Drug: Tolcapone; Drug: Placebo

INTERVENTIONS:
Drug: Tolcapone — Tolcapone 100 mg tablets
  Other Names: Tasmar
Drug: Placebo — Placebo tablets

SUMMARY:
The purpose of this study is to determine whether the catechol-O-methyltransferase (COMT) inhibitor tolcapone, relative to placebo, affects response to alcohol, decision-making, brain activation associated with alcohol cue reactivity, response inhibition, and selective attention, or alcohol drinking.

DETAILED DESCRIPTION:
This study evaluates the effects of an FDA-approved medication called tolcapone in people who have both Alcohol Use Disorder (AUD) and Attention-Deficit/Hyperactivity Disorder (ADHD). The study involves seven visits over a three to four week period, including an assessment visit and two eight-day medication periods during which participants will be assigned to take, in a double-blinded fashion, both tolcapone and a placebo (three visits during each period). During two of these visits, participants will undergo a one-hour MRI scan. Participants must not be seeking treatment for AUD or ADHD and must not be currently taking any psychotropic medications, including stimulant medications for ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65.
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current Alcohol Use Disorder (AUD) and current Attention-Deficit/Hyperactivity Disorder (ADHD), as assessed by the Structured Clinical Interview for DSM-5 (SCID-5) or WHO-ASRS.
3. Currently not engaged in, and does not want treatment for, AUD or ADHD.
4. Currently not taking any medication for AUD or ADHD.
5. Able to read and understand questionnaires and informed consent.
6. Lives within 50 miles of the study site.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
2. Any psychoactive substance use (except nicotine) within the last 30 days, as indicated by self-report and urine drug screen (UDS)
3. Current DSM-5 psychotic, mood, anxiety, obsessive-compulsive, trauma-related, or eating disorder, as assessed by SCID-5.
4. Current suicidal ideation or homicidal ideation.
5. Current use of any psychoactive medication, as evidenced by self-report and UDS.
6. History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self-report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
7. Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems, as evidenced by medical history and physical exam.
8. Past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, or peptic ulcer.
9. Current or past hepatocellular disease, as indicated by verbal report, or elevations of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than the upper limit of the normal range at screening.
10. Females of childbearing potential who are pregnant (by plasma HCG), nursing, or who are not using a reliable form of contraception.
11. Current charges pending for a violent crime (not including DUI-related offenses).
12. Lack of a stable living situation.
13. Presence of ferrous metal in the body, as evidenced by metal screening and self-report.
14. Severe claustrophobia or morbid obesity that preclude placement in the MRI scanner.
15. History of neurological disease or head injury with > 2 minutes of unconsciousness.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol-induced stimulation between medication periods | 30 minutes after laboratory alcohol administration on Day 1 of each medication period. Each medication period is 8 days long.
  Biphasic Alcohol Effects Scale stimulation score (range = 0-70; higher scores = more stimulation) after laboratory alcohol administration
Change in subjective response to alcohol between medication periods | 30 minutes after laboratory alcohol administration on Day 1 of each medication period. Each medication period is 8 days long.
  Subjective High Assessment Scale (range - 0-130; higher scores = greater intoxication) after laboratory alcohol administration
Change in risky decision-making after alcohol administration between medication periods | 30 minutes after laboratory alcohol administration on Day 1 of each medication period. Each medication period is 8 days long.
  Balloon Analogue Risk Task adjusted average number of pumps (higher scores = more risky decision-making)
Change in cognitive-control-associated brain activation (fMRI) between medication periods | 60 minutes after medication ingestion on Day 2 of each medication period. Each medication period is 8 days long.
  Stop-signal task blood oxygenation level dependent (BOLD) signal to successful stop trials, relative to unsuccessful stop trials
Change in selective attention-associated brain activation (fMRI) between medication periods | 60 minutes after medication ingestion on Day 2 of each medication period. Each medication period is 8 days long.
  Multi-source interference task BOLD signal to interference trials, relative to control trials
Change in alcohol cue-elicited brain activation (fMRI) between medication periods | 60 minutes after medication ingestion on Day 2 of each medication period. Each medication period is 8 days long.
  Alcohol cue reactivity task BOLD signal to alcohol cues, relative to neutral beverage cues

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Schacht, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No